CLINICAL TRIAL: NCT02365116
Title: Peer Mentorship to Reduce Suicide Risk Following Psychiatric Hospitalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Paul Pfeiffer, Assistant Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH103447-01 (NIH)
Record Dates: First submitted 2014-05-28; First posted 2015-02-18 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Suicidal Ideation
Keywords: Peer Mentorship; Psychiatric Hospitalization; Suicide Risk
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peer Mentorship intervention (Experimental): A Peer Specialist will be making weekly follow-up contact with study participants in the community or by telephone for 3 months following hospital discharge. The content of the peer mentorship interactions will be based on the manual developed by the study team and will include components such as hope and belongingness.
  Interventions: Behavioral: Peer mentorship
- Enhanced Usual Care (Active Comparator): Patients will continue to receive usual care which typically consists of referral to an outpatient psychiatrist. Participants will also receive a phone call within 24-72 hours from a member of the inpatient unit clinical staff to assess barriers to follow-up care and safety. The enhancement to usual care will occur at the 3 and 6 month follow-up assessments, where participants will be assessed to determine whether they require any additional referral information for follow-up care. If referral information is indicated, the patient will be provided a list of mental health treatment providers in their area.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Peer mentorship — Patients who are working with a peer specialist will have their sessions audio taped and reviewed by research staff for training purposes and to ensure that peer specialists are following protocol.
  Arms: Peer Mentorship intervention
Behavioral: Enhanced Usual Care — The enhancement to usual care will occur at the 3 and 6 month follow-up assessments, where participants will be assessed to determine whether they require any additional referral information for follow-up care. If referral information is indicated, the patient will be provided a list of mental health treatment providers in their area.
  Arms: Enhanced Usual Care

SUMMARY:
Every year in the United States about 1 million people make a suicide attempt and more than 38,000 die by suicide. The risk of suicide is highest among individuals with mental illness who have been hospitalized due to suicidal thoughts or behaviors, yet there are few interventions known to reduce suicide risk in this population. This study will develop and pilot test a peer mentorship intervention by which trained peer professionals will use their own personal experience with recovery from mental illness to instill hope and belongingness in high-risk patients and provide additional support to prevent future suicidal thoughts or behaviors.

The specific aims of the study are to: (1) develop a peer mentorship intervention to reduce suicide risk among patients psychiatrically hospitalized with suicidal ideation or following a suicide attempt; (2) Conduct a randomized controlled pilot study to assess the acceptability, feasibility, and fidelity of the peer mentorship intervention in preparation for a larger efficacy trial; and (3) an exploratory aim will be to measure potential mediators and moderators of intervention effectiveness in terms of belongingness, burdensomeness, and hopelessness according to the interpersonal theory of suicide.

ELIGIBILITY:
Inclusion Criteria:

1. are age 18 years or older
2. have medical record documentation of suicidal ideation or suicide attempt at the time of admission
3. are fluent in English

Exclusion Criteria:

1. substantially cognitively impaired (according to Mini-Cog)
2. unable to provide voluntary, written, informed consent for any reason (including incompetency)
3. determined by the patient's attending psychiatrist that due to the patient's psychiatric condition peer mentorship may be harmful to the patient or peer specialist (e.g., severe personality disorder, unstable paranoia)
4. already receiving or intending to receive peer mentorship (including having a sponsor from Alcoholics Anonymous) or participate in group-based peer support on a biweekly or more frequent basis
5. are receiving electroconvulsive therapy (ECT)
6. are located more than 50 miles from any of the peer specialists
7. are being discharged to a residential treatment facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-08-19 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-26 (Actual)

PRIMARY OUTCOMES:
Intervention acceptability (median number of peer mentorship contacts at 3 months post-discharge is at least 4, as well as by satisfaction questionnaires.) | 3 and 6 months post-baseline
  Patients' willingness and satisfaction with participating in the intervention as a measure of intervention acceptability. Measured by at least 70% of participants in both study arms completing follow-up measures at 6 months, the median number of peer mentorship contacts at 3 months post-discharge is at least 4, as well as by satisfaction questionnaires.
Intervention feasibility (Study team's ability to deliver the intervention) | 3 and 6 months post-baseline
  Study team's ability to deliver the intervention as a measure of feasibility. Measured by at least 50% of eligible patients choosing to enroll in the study, at least 80% of participants assigned to the peer mentorship arm meeting with a peer specialist prior to hospital discharge, at least 70% of participants in both study arms completing follow-up measures at 6 months, and the study meeting its enrollment goal of 60 patients in 12 months.

SECONDARY OUTCOMES:
Current suicidal ideation (measured by the Beck Suicide Scale (BSS) | 3 and 6 months post-baseline
  Patient's current suicidal ideation as measured by the Beck Suicide Scale (BSS)
Peak suicidal ideation (measured by the Columbia Suicide Severity Rating Scale (CSSR-S) | 3 and 6 months post-baseline
  Patient's peak suicidal ideation since the last visit as measured by the Columbia Suicide Severity Rating Scale (CSSR-S)
Suicide attempts (measured by the Columbia Suicide Severity Rating Scale) | 3 and 6 months post-baseline
  Patient's suicide attempts since the last visit as measured by the Columbia Suicide Severity Rating Scale

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Michigan Inpatient Psychiatry Unit, Ann Arbor, Michigan
  - Henry Ford Kingswood Hospital, Ferndale, Michigan

IPD SHARING:
Plan to Share IPD: No